CLINICAL TRIAL: NCT01806675
Title: Phase 1-2 18F-FPPRGD2 PET/CT or PET/MRI Imaging of αvβ3 Integrins Expression as a Biomarker of Angiogenesis
Brief Title: 18F-FPPRGD2 PET/CT or PET/MRI in Predicting Early Response in Patients With Cancer Receiving Anti-Angiogenesis Therapy
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sanjiv Sam Gambhir (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, Sanjiv Sam Gambhir, Virginia and D.K. Ludwig Professor for Clinical Investigation in Cancer Research, Stanford University
Organization: Stanford University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB-25970; NCI-2013-00535 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); IRB-25970 (Other: Stanford IRB); VARIMG0002 (Other: OnCore ID)
Record Dates: First submitted 2013-03-05; First posted 2013-03-07 (Estimated); Results first posted 2019-09-06 (Actual); Last update posted 2019-10-03 (Actual); Status verified 2019-09

CONDITIONS: Adult Giant Cell Glioblastoma; Adult Glioblastoma; Adult Gliosarcoma; Male Breast Cancer; Metastatic Squamous Neck Cancer With Occult Primary Squamous Cell Carcinoma; Recurrent Adenoid Cystic Carcinoma of the Oral Cavity; Recurrent Adult Brain Tumor; Recurrent Basal Cell Carcinoma of the Lip; Recurrent Colon Cancer; Recurrent Esthesioneuroblastoma of the Paranasal Sinus and Nasal Cavity; Recurrent Hypopharyngeal Cancer; Recurrent Inverted Papilloma of the Paranasal Sinus and Nasal Cavity; Recurrent Laryngeal Cancer; Recurrent Lip and Oral Cavity Cancer; Recurrent Lymphoepithelioma of the Nasopharynx; Recurrent Lymphoepithelioma of the Oropharynx; Recurrent Metastatic Squamous Neck Cancer With Occult Primary; Recurrent Midline Lethal Granuloma of the Paranasal Sinus and Nasal Cavity; Recurrent Mucoepidermoid Carcinoma of the Oral Cavity; Recurrent Nasopharyngeal Cancer; Recurrent Non-small Cell Lung Cancer; Recurrent Oropharyngeal Cancer; Recurrent Pancreatic Cancer; Recurrent Paranasal Sinus and Nasal Cavity Cancer; Recurrent Rectal Cancer; Recurrent Renal Cell Cancer; Recurrent Salivary Gland Cancer; Stage IIIA Breast Cancer; Stage IIIA Non-small Cell Lung Cancer; Stage IIIB Breast Cancer; Stage IIIB Non-small Cell Lung Cancer; Stage IIIC Breast Cancer; Stage IV Breast Cancer; Stage IV Non-small Cell Lung Cancer; Stage IV Pancreatic Cancer; Stage IV Renal Cell Cancer; Stage IVA Colon Cancer; Stage IVA Rectal Cancer; Stage IVA Salivary Gland Cancer; Stage IVB Colon Cancer; Stage IVB Salivary Gland Cancer; Stage IVC Salivary Gland Cancer; Tongue Cancer; Unspecified Adult Solid Tumor, Protocol Specific
MeSH Terms: conditions — Glioblastoma; Gliosarcoma; Breast Neoplasms, Male; Brain Neoplasms; Colonic Neoplasms; Esthesioneuroblastoma, Olfactory; Hypopharyngeal Neoplasms; Laryngeal Neoplasms; Mouth Neoplasms; Nasopharyngeal Neoplasms; Carcinoma, Non-Small-Cell Lung; Oropharyngeal Neoplasms; Pancreatic Neoplasms; Rectal Neoplasms; Carcinoma, Renal Cell; Salivary Gland Neoplasms; Breast Neoplasms; Tongue Neoplasms | interventions — Fluorodeoxyglucose F18; FPP(RGD)2

STUDY DESIGN:
Masking Description: All human subject participants were to be evaluated with both 18F-FPPRGD2 PET/CT and 18-FDG PET/CT imaging scans.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Glioblastoma Multiforme (GBM) (Experimental): Patients with glioblastoma multiforme (GBM) undergo 18F-FDG and 18F-FPPRGD2 positron emission tomography / computed tomography (PET/CT) imaging at baseline and 6 weeks (or standard of care follow-up)
  Interventions: Drug: 18F-fludeoxyglucose (18F-FDG); Drug: 18F-FPPRGD2
- Gynecological Cancers (Experimental): Patients with gynecological cancer undergo 18F-FDG and 18F-FPPRGD2 positron emission tomography / computed tomography (PET/CT) imaging at baseline and at 9 t0 12 weeks (or standard of care follow-up)
  Interventions: Drug: 18F-fludeoxyglucose (18F-FDG); Drug: 18F-FPPRGD2
- Renal Cell Cancer (RCC) (Experimental): Patients with renal cell cancer (RCC) undergo 18F-FDG and 18F-FPPRGD2 positron emission tomography / computed tomography (PET/CT) imaging at baseline and at 9 t0 12 weeks (or standard of care follow-up)
  Interventions: Drug: 18F-fludeoxyglucose (18F-FDG); Drug: 18F-FPPRGD2

INTERVENTIONS:
Drug: 18F-fludeoxyglucose (18F-FDG) — 18F-FDG will be used as the radiotracer for a regular medical care PET/CT or PET/MRI scan
  Other Names: Fludeoxyglucose F-18; 18-FDG; FDG
Drug: 18F-FPPRGD2 — 18F-FPPRGD2 will be used as the radiotracer for a PET/CT or PET/MRI scan. Participants will be injected with less than 10 mCi of 18F-FPPRGD2.
  Other Names: (18F)-2-fluoropropionyl-labeled PEGylated dimeric arginine-glycine-aspartic acid peptide; [PEG3-E{c(RGDyk)}2]; fluorine-18-FPPRGD2; [18F]-FPPRGD2; 2-fluoropropionyl-labeled pegylated dimeric RGD peptide; 104150

SUMMARY:
The purpose of the study is to conduct research of a new PET radiopharmaceutical in cancer patients. The uptake of the novel radiopharmaceutical 18F-FPPRGD2 will be assessed in study participants with glioblastoma multiforme (GBM), gynecological cancers, and renal cell carcinoma (RCC) who are receiving antiangiogenesis treatment.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE

• Evaluate 18F-FPPRGD2 and 18F-FDG as PET/CT or PET/MRI radiotracers for imaging prediction and assessment of response to anti-angiogenesis therapy in participants with glioblastoma multiforme (GBM), gynecological cancers, and renal cell carcinoma (RCC).

SECONDARY OBJECTIVE

• Progression-free survival (PFS) at up to 1 year after initial scans and treatment

OUTLINE:

Patients undergo 18F-FPPRGD2 and 18F-FDG PET/CT or PET/MRI medical imaging at baseline and at regular medical care follow-up (6 to 12 weeks).

After completion of study imaging, patients are followed up at 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Provides written informed consent
* Diagnosed with advanced NSCLC, breast cancer, GBM or other cancers (such as head and neck, colorectal, pancreatic, renal cancers); patients will undergo anti-angiogenesis treatment or treatment with other drugs that may alter angiogenesis
* Able to remain still for duration of each imaging procedure (about one hour)

Exclusion Criteria:

* Pregnant or nursing
* Contraindication to MRI
* History of renal insufficiency (only for MRI contrast administration)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2013-03-04 (Actual); Primary Completion 2016-12-07 (Actual); Study Completion 2019-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sanjiv Gambhir, MD, PhD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, School of Medicine, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Minamimoto R, Jamali M, Barkhodari A, Mosci C, Mittra E, Shen B, Chin F, Gambhir SS, Iagaru A. Biodistribution of the (1)(8)F-FPPRGD(2) PET radiopharmaceutical in cancer patients: an atlas of SUV measurements. Eur J Nucl Med Mol Imaging. 2015 Nov;42(12):1850-8. doi: 10.1007/s00259-015-3096-4. Epub 2015 Jun 11. PMID 26062933
- [Result] Iagaru A, Mosci C, Mittra E, Zaharchuk G, Fischbein N, Harsh G, Li G, Nagpal S, Recht L, Gambhir SS. Glioblastoma Multiforme Recurrence: An Exploratory Study of (18)F FPPRGD2 PET/CT. Radiology. 2015 Nov;277(2):497-506. doi: 10.1148/radiol.2015141550. Epub 2015 May 12. PMID 25965900
- [Result] Minamimoto R, Karam A, Jamali M, Barkhodari A, Gambhir SS, Dorigo O, Iagaru A. Pilot prospective evaluation of (18)F-FPPRGD2 PET/CT in patients with cervical and ovarian cancer. Eur J Nucl Med Mol Imaging. 2016 Jun;43(6):1047-55. doi: 10.1007/s00259-015-3263-7. Epub 2015 Nov 27. PMID 26611425
- [Result] Toriihara A, Duan H, Thompson HM, Park S, Hatami N, Baratto L, Fan AC, Iagaru A. 18F-FPPRGD2 PET/CT in patients with metastatic renal cell cancer. Eur J Nucl Med Mol Imaging. 2019 Jul;46(7):1518-1523. doi: 10.1007/s00259-019-04295-7. Epub 2019 Mar 8. PMID 30850872

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Glioblastoma Multiforme (GBM) | Gynecological Cancers | Renal Cell Cancer (RCC)
Started | 11 | 6 | 8
Completed | 11 | 6 | 8
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Glioblastoma Multiforme (GBM) | Gynecological Cancers | Renal Cell Cancer (RCC) | Total
Number analyzed (Participants) | 11 | 6 | 8 | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 11 | 6 | 4 | 21
  >=65 years | 0 | 0 | 4 | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.1 (8.3) | 44.3 (12.6) | 64.1 (13.3) | 54.9 (13.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 6 | 3 | 14
  Male | 6 | 0 | 5 | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 1 | 3
  Not Hispanic or Latino | 10 | 5 | 7 | 22
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 2 | 3 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 8 | 2 | 4 | 14
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 2 | 2 | 1 | 5
Region of Enrollment [Number; unit: participants]
  United States | 11 | 6 | 8 | 25

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Maximum Standard Uptake Values (SUVmax)
Description: Maximum standard uptake values (SUVmax) were assessed on the basis of position emission tomography (PET) scans using radiotracers 18F-FPPRGD2 and 18F-FDG at baseline and at regular medical care follow-up (6 to 12 weeks after initiation of treatment). The outcome is assessed as the difference in the maximum standard uptake values (SUVmax) values from baseline to follow-up for the 2 radiotracers, and will be reported for each disease type as the median with standard deviation.
Time Frame: At baseline and 6 weeks
Population: Some participants did not contribute some or all post-treatment scans.
Measure: Median (Standard Deviation); unit: ratio
Arm/Group | Glioblastoma Multiforme (GBM) | Gynecological Cancers | Renal Cell Cancer (RCC)
Number analyzed (Participants) | 8 | 4 | 4
ratio
  18F-FPPRGD2 PET scans: number analyzed (Participants) | 8 | 4 | 3
  18F-FPPRGD2 PET scans | -0.98 (0.98) | 0.09 (1.20) | 0.10 (0.29)
  18F-FDG PET scans: number analyzed (Participants) | 0 | 4 | 3
  18F-FDG PET scans |  | -1.90 (2.80) | 7.8 (8.2)

2. Secondary Outcome: Response Assessment by RANO Criteria
Description: The treatment effect for participants with glioblastoma multiforme was to be assessed on the basis of post-treatment evaluation per the Response Assessment in Neuro-Oncology (RANO) Criteria. The outcome was the number & proportion of participants that achieved either a complete response (CR) or partial response (PR), a number without dispersion. RANO criteria are:
  CR= No T1 gadolinium (T1-G); T2-weighted-Fluid-Attenuated Inversion Recovery (T2/FLAIR) stable/decreased, no new lesions; no corticosteroids; clinical condition improved/stable.
  PR= ≥50% decrease in T1-G; T2/FLAIR decreased/stable ; no new lesions; decreased/stable corticosteroids; clinical condition improved/stable.
  Stable disease (SD)= <50% decrease, but more than 25% increase, in T1-G; T2/FLAIR decreased/stable; no new lesions; decreased/stable corticosteroids; clinical condition improved/stable.
  Progressive disease (PD)= ≥25%increase T1-G; T2/FLAIR increased; increased corticosteroids; clinical condition decreased
Time Frame: At baseline and 6 weeks
Population: This assessment was restricted to glioblastoma multiforme (GBM) participants only, however, no response assessments were obtained for GBM participants.
Arm/Group | Glioblastoma Multiforme (GBM) | Gynecological Cancers | Renal Cell Cancer (RCC)
Number analyzed (Participants) | 0 | 0 | 0

3. Secondary Outcome: Change in Tumor Size
Description: The treatment effect for participants with gynecological cancers (GYN) and renal cell carcinoma (RCC) was assessed on the basis of change in tumor size as determined by pre- and post-treatment CT scans. The outcome is reported as the difference at treatment follow-up, reported as the median with standard deviation.
Time Frame: 9 to 12 weeks
Population: This assessment was restricted to gynecological cancers and renal cell carcinoma participants only. Tumor response data was not available for all participants in these groups.
Measure: Median (Standard Deviation); unit: centimeters
Arm/Group | Glioblastoma Multiforme (GBM) | Gynecological Cancers | Renal Cell Cancer (RCC)
Number analyzed (Participants) | 0 | 3 | 3
centimeters |  | 0.9 (1.56) | 1 (1.56)

4. Secondary Outcome: Tumor Response Rate by EORTC Criteria
Description: Tumor Response Rate by EORTC Criteria Tumor response rates were assessed from position emission tomography (PET) scans using 18F-FPPRGD2 & 18F-FDG at baseline & after 6 weeks of treatment, per European Organization for Research & Treatment of Cancer (EORTC) response criteria. The outcome is reported for each radiotracer by disease group as the number of participants achieving complete response (CR), partial response (PR), stable disease (SD), & progressive disease (PD).
  * CR= complete resolution of 18F-FDG uptake tumor volume
  * PR= reduction of 15-25% in tumor 18F-FDG SUVmax after 1 cycle of chemotherapy, and ≥25% after >1 cycle
  * SD= increase in tumor 18F-FDG SUVmax of <25% or a decrease of <15% & no increase in 18F-FDG tumor uptake [>20% in the longest dimension (LD)];
  * PD= increase in 18F-FDG tumor SUVmax of >25% in tumor region on baseline; increase in extent of 18F-FDG tumor uptake (>20% in LD); appearance of new 18F-FDG uptake in metastatic lesions
Time Frame: At baseline and 6 weeks
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | Glioblastoma Multiforme (GBM) | Gynecological Cancers | Renal Cell Cancer (RCC)
Number analyzed (Participants) | 0 | 4 | 4
participants
  Complete Response (CR) |  | 2 | 0
  Partial Repsonse (PR) |  | 1 | 0
  Stable Disease (SD) |  | 0 | 2
  Progressive Disease |  | 1 | 2

5. Secondary Outcome: Progression-free Survival (PFS)
Description: Progression-free survival (PFS) was defined as remaining alive at 1 year with disease progression, according to the physician's assessment of clinical status, by disease group.
Time Frame: 1 year
Population: Data was not collected for progression-free survival (PFS).
Arm/Group | Glioblastoma Multiforme (GBM) | Gynecological Cancers | Renal Cell Cancer (RCC)
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: 6 weeks
Arm/Group | Glioblastoma Multiforme (GBM) | Gynecological Cancers | Renal Cell Cancer (RCC)
All-Cause Mortality (participants affected / at risk) | 1/11 | 0/6 | 0/8
Serious Adverse Events (participants affected / at risk) | 1/11 | 0/6 | 2/8
Other Adverse Events (participants affected / at risk) | 0/11 | 0/6 | 0/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Glioblastoma Multiforme (GBM) (N=11) | Gynecological Cancers (N=6) | Renal Cell Cancer (RCC) (N=8)
Death NOS (General disorders) | 1 (1) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes